CLINICAL TRIAL: NCT05830318
Title: Usability and Acceptability Study of the P-STEP Mobile Application
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Leicester (Other)
Responsible Party: Sponsor
Other Study IDs: 0901
Record Dates: First submitted 2023-03-16; First posted 2023-04-26 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-07

CONDITIONS: Asthma; Chronic Obstructive Pulmonary Disease; Interstitial Lung Disease; Coronary Heart Disease; Heart Failure; Type 2 Diabetes
Keywords: Exercise; Pollution; Air Quality
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive; Lung Diseases, Interstitial; Coronary Disease; Heart Failure; Diabetes Mellitus, Type 2; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: P-STEP Mobile Application — A mobile application that allows you track your walking habits while keeping you up to date with air quality information.

SUMMARY:
Assess the usability and acceptance of the P-STEP app, through allowing participants with specific chronic conditions to pilot the app for 12-weeks.

DETAILED DESCRIPTION:
Participants are asked to use mobile app for 12 weeks & complete baseline, 6 week and 12 week assessments.

ELIGIBILITY:
Inclusion Criteria:

* Adult ≥ 18 years
* Live within the boundaries of the test site (Leicester, UK).
* Diagnosed with one (or more) of the following conditions: asthma, chronic obstructive pulmonary disease (COPD), interstitial lung disease (ILD), coronary heart disease (CHD), heart failure (HF), type 2 diabetes
* Android smartphone which has access to the internet
* Can walk outside for a minimum of 5 minutes without feeling uneasy/unsteady
* Available to pilot the app for 12 weeks from August-December 2023
* Able to give informed consent to participate in the evaluation

Exclusion Criteria:

* English language restriction
* Advised not to do exercise by a health care professional, in the last 12 months.
* Access to an iOS smartphone only
* Diagnosed with dementia, learning disability, mental health disorders (other than depression or anxiety), epilepsy
* Receiving palliative care
* Pregnant
* Chest pain at rest
* Unsteady when standing or walking
* Current cancer patient
* Part of the P-STEP User Engagement group

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential participants will be identified and recruited on a voluntary basis exclusively from the EXCEED cohort study. A longitudinal cohort study based in Leicester, UK.
Sampling Method: Non-Probability Sample
Enrollment: 380 (Estimated)
Dates: Start 2023-08-23 (Actual); Primary Completion 2023-12-22 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
System Usability Scale | 12 weeks
  the System Usability Scale (SUS) at 12 weeks. The SUS a validated scale and a popular instrument for assessing perceived usability. There are 10 items in total, 5 with a positive tone and 5 with a negative tone, the response of each ranging from strongly disagree to strongly agree. The participant's scores will be transformed onto a 0-100 scale. General guidance suggests a SUS score 68 and above to be considered above average and below 68 is below average. Scores range from 0-100, a higher score indicates higher usability.

SECONDARY OUTCOMES:
Usability of P-STEP app | 12 weeks
  Other than the SUS, 9 usability questions relating to the specific features of the app will be asked. Participants will also be asked to provide their general feedback on the app as well as how much they used it. Individual items in the questionnaire will be summarised with percentages. Scores range from 1-5, a higher score indicates higher usability.
User Engagement Scale Short Form | 12 weeks
  The User Engagement Scale - Short Form (UES-SF) is a reliable a valid questionnaire containing twelve items that measure user engagement categorised into; focused attention, perceived usability, aesthetic appeal, and reward. These categories can be calculated to get an average of the scores. An overall user engagement score can be calculated with UES-SF by adding together all 12 items and dividing them equally. Scores are presented on a scale 1-5. The items can be averaged into 4 categories or averaged for an overall score. Scores range from 0-60, a higher score indicates higher user engagement.
SF-12 Health Questionnaire | 12 weeks
  The short form 12 item (SF-12v2) health survey measures functional health and well-being from the participant's perspective. It assesses eight domains; physical functioning, physical role, pain, general health, vitality, social functioning, social role, mental health. Each domain contributes to two summary scores; physical component summary (PCS) and mental component summary (MCS). SF-12v2 responses will be scored and interpreted using the SF-12v2 user guide. The 8 domains will generate two summary scores; physical component score (PCS) and mental component score (MCS). Scores for the PCS and MCS range from 0-100, a higher score indicates a higher quality of life.
Recent Physical Activity Questionnaire | 12 weeks
  The RPAQ is designed to find out about a participant's physical activity in their everyday life. The RPAQ will be scored and interpreted using the scoring guidelines published by the Authors. All activities are categorised with respect to their intensity, on a scale of sedentary (<1.5), light (1.5-<3), moderate (3-6) and vigorous (>6). Each activity is scored by hours a day multiplied by the intensity of the activity. A higher RPAQ score indicates higher levels of physical activity.
Feasibility outcome - Interest | 2 months
  Percentage of those potentially eligible who register their interest.
Feasibility outcome - Enrolment | 2 months
  Percentage of participants that register interest enrol on the study.
Feasibility outcome - App administration | 3 months
  Percentage that successfully download the app.
Feasibility outcome - App acceptability | 3 months
  Percentage of participants who enrol and complete the 12-week study
Feasibility outcome - Acceptability of the outcome measures | 3 months
  Completion levels of questionnaire
All cause mortality | 3 months
  Description of all cause mortality at 3 months
Cardiovascular events | 3 months
  Description of cardiovascular events at 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Leicester, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Worboys HM, Gray LJ, Anthony S, Hobson R, Lucas T, Vande Hey JD, Panagi M, Ng GA. A feasibility study evaluating the usability and acceptability of the personalised space technology exercise platform mobile application. Sci Rep. 2025 Oct 17;15(1):36370. doi: 10.1038/s41598-025-20314-0. PMID 41107355
- [Derived] Worboys H, Gray L, Anthony S, Hobson R, Lucas T, Ng A. Evaluation of the usability and acceptability of the P-STEP(R) mobile app: feasibility study protocol. Pilot Feasibility Stud. 2024 Sep 13;10(1):120. doi: 10.1186/s40814-024-01546-9. PMID 39272125